CLINICAL TRIAL: NCT06100666
Title: Investigation of Sustainable Eating Behaviors and Diet Quality in Adults
Brief Title: Sustainable Eating Behaviors and Diet Quality
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Tarsus University (Other)
Responsible Party: Principal Investigator, Gamze Altıntaş, Principal Investigator, Ankara University
Other Study IDs: AU-BES-GAltintas-001
Record Dates: First submitted 2023-10-15; First posted 2023-10-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Nutrition, Healthy
Keywords: Anthropometry; Diet, Food, and Nutrition; Diet Records; Eating; Health Behavior; Nutrition Assessment; Sustainable Development
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Academic and administrative staff working at Tarsus University
  Interventions: Behavioral: Observational Tests

INTERVENTIONS:
Behavioral: Observational Tests — The Sustainable and Healthy Eating Behaviors Scale will be used to assess sustainable eating behaviors, one-day food consumption records will be collected with the 24-hour Dietary Recall method, the International Diet Quality Index and EAT-Lancet Diet Score will be used to assess diet quality, and body weight, height, waist circumference and neck circumference will be measured to determine nutritional status.

SUMMARY:
The goal of this observational study is to evaluate the sustainable nutrition behaviors (e.g. not wasting food, consuming organic food) and diet quality of university staff. The main questions it aims to answer are:

* What is the diet quality of the participants?
* Do participants with higher diet quality have better sustainable eating behaviors?

DETAILED DESCRIPTION:
Sustainable diets are diets with low environmental impacts that contribute to food and nutritional security and healthy living for present and future generations. They are recognized as protective of ecosystems, culturally acceptable, accessible, economically fair and affordable, nutritionally adequate, safe and healthy diets. Sustainable healthy diets ensure optimal growth and development of all individuals, support functionality across all life stages for current and future generations, contribute to the prevention of all forms of malnutrition, reduce the risk of diet-related non-communicable diseases and support the protection of biodiversity and planetary health. Recently, the need to promote nutritious and safe sustainable diets with low environmental impact has been emphasized. Diets based mostly on plant-based foods, such as the Mediterranean diet and the DASH diet, are recognized as sustainable eating models. The aim of this study is to evaluate the sustainable eating behaviors and diet quality based on food consumption of academic and administrative staff working at the university and to determine the relationship between them.

1. How is the diet quality of the university staff?
2. How are the sustainable nutrition behaviors of the university staff?
3. Is there a difference between diet quality groups in terms of sustainable nutrition behaviors?

ELIGIBILITY:
Inclusion Criteria:

* Being a staff member of Tarsus University
* Volunteering to participate in the study

Exclusion Criteria:

* Pregnancy
* The presence of any known condition that prevents the taking of anthropometric measurements
* Presence of a known memory problem that may prevent receiving 24-hour Recall

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tarsus University academic and administrative staff
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
24-hour Dietary Recall | 1 year
  To assess the diet quality of the participants. It will be evaluated using the Nutrition Information System (BeBiS). In the 24-hour Dietary Recall, the foods consumed at all meals, the contents and quantities of the meals will be questioned. Standard recipes will be used for foods or meals consumed outside the home.
Sustainable and Healthy Eating Behaviors Scale | 1 year
  It will be used to assess participants' sustainable nutrition behaviors. The Turkish version of the scale consists of 7 factors and 32 Likert-type questions, including Quality Marks (Local and Organic), Seasonal Foods and Avoiding Food Waste, Animal Health, Reducing Meat Consumption, Healthy and Balanced Nutrition, Local Food and Low Fat. Respondents are asked to rate the questions as never, very rarely, rarely, sometimes, often, very often and always. Never=1 point and Always=7 points. There is no intercept value in the evaluation, a high score indicates an increase in sustainable and healthy eating behavior.
International Diet Quality Index | 1 year
  To be used to assess diet quality. This index was developed to assess and compare diet quality across countries. It assesses four components of the diet: variety, adequacy, moderation and overall balance. The sum of the scores in these four main categories determines the total score for the index. The total score ranges from 0-100 (0= lowest diet quality, 100= highest diet quality). According to the index total score, a score of 0- ≤45 points is classified as poor diet quality, >55- ≤60 points as moderate diet quality, and >75 points as high diet quality.
Body weight in kilograms | 1 year
  Body weight measurement will be made with a weighing device sensitive to 0.5 kg.
Height in meters | 1 year
  A stadiometer will be used to measure height and measurements will be recorded with an accuracy of 0.1 cm. The measurement will be made without shoes, feet together, head in the Frankfurt plane, and head, back, hips, calves and heels in the same plane.
Waist circumference in centimeters | 1 year
  Waist circumference will be measured at the midpoint between the lowest rib and the iliac crest using a non-stretchable tape measure. The measurement will be repeated twice and averaged.
Neck circumference in centimeters | 1 year
  Neck circumference will be measured in the middle of the neck, between the mid-cervical spine and mid-anterior neck, using a non-stretchable tape measure while the participants are standing upright, and recorded with an accuracy of 0.1 cm. In men with a laryngeal protrusion, it will be measured just below the protrusion.

SECONDARY OUTCOMES:
EAT-Lancet Diet Score | 1 year
  It includes 14 main recommendations. For different food groups, a score of "1" is given if the person consumed the specified amount and a score of "0" if the person did not consume the specified amount. The maximum score for this diet score is 14.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Altintas, Principal Investigator — Ankara University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- [Background] Hanley-Cook GT, Argaw AA, de Kok BP, Vanslambrouck KW, Toe LC, Kolsteren PW, Jones AD, Lachat CK. EAT-Lancet diet score requires minimum intake values to predict higher micronutrient adequacy of diets in rural women of reproductive age from five low- and middle-income countries. Br J Nutr. 2021 Jul 14;126(1):92-100. doi: 10.1017/S0007114520003864. Epub 2020 Sep 30. PMID 32993824
- [Background] Kim S, Haines PS, Siega-Riz AM, Popkin BM. The Diet Quality Index-International (DQI-I) provides an effective tool for cross-national comparison of diet quality as illustrated by China and the United States. J Nutr. 2003 Nov;133(11):3476-84. doi: 10.1093/jn/133.11.3476. PMID 14608061
- [Background] Knuppel A, Papier K, Key TJ, Travis RC. EAT-Lancet score and major health outcomes: the EPIC-Oxford study. Lancet. 2019 Jul 20;394(10194):213-214. doi: 10.1016/S0140-6736(19)31236-X. Epub 2019 Jun 21. No abstract available. PMID 31235280
- [Background] Koksal E, Bilici S, Citar Daziroglu ME, Erdogan Govez N. Validity and Reliability of the Turkish Version of the Sustainable and Healthy Eating Behaviors Scale. Br J Nutr. 2022 Aug 8:1-20. doi: 10.1017/S0007114522002525. Online ahead of print. PMID 35938236
- [Background] Zakowska-Biemans S, Pieniak Z, Kostyra E, Gutkowska K. Searching for a Measure Integrating Sustainable and Healthy Eating Behaviors. Nutrients. 2019 Jan 5;11(1):95. doi: 10.3390/nu11010095. PMID 30621258
- [Derived] Altintas-Mutlu G, Ucar A. Assessment of sustainable and healthy eating behaviors, EAT-lancet diet score, diet quality and obesity indicators among university staff: a cross-sectional study. J Health Popul Nutr. 2025 Nov 12;44(1):397. doi: 10.1186/s41043-025-01124-6. PMID 41225681